CLINICAL TRIAL: NCT07018687
Title: Improvement of Nutritional Status in Cancer Patients and Reduction of Malnutrition
Acronym: NUTRI-CARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Médipôle Lyon-Villeurbanne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NUTRI-CARE
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Patient Readmission

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Dietician consultation
  Interventions: Other: dietician consultation
- day hospital (Experimental): mutlidisciplinary care
  Interventions: Other: day hospital

INTERVENTIONS:
Other: day hospital — This multidisciplinary day hospital consists of 3 information workshops focused on balanced nutrition, oral nutritional supplements and enrichments as well as artificial feeding. During this day hospital, patients will meet with an endocrinologist nutritionist, a dietitian, and a teacher in adapted physical activity.
  Arms: day hospital
Other: dietician consultation — dietician consultation
  Arms: Control

SUMMARY:
The European Society for Clinical Nutrition and Metabolism (ESPEN) recommends assessing the nutritional status of each oncology patient early and in a multidisciplinary manner.

This assessment should take into account physical activity and should allow for the patient to be provided with nutritional goals adapted to their new needs. These recommendations aim to combat malnutrition, which sometimes leads to treatment suspension and thus a loss of opportunity for the patient.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed cancer

Exclusion Criteria:

* other cancer previously diagnosed
* under 18 years old
* pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2026-04-08 (Estimated)

PRIMARY OUTCOMES:
weight loss | 1 year

SECONDARY OUTCOMES:
quality of life sf-36 | 1 year
  sf-36

CONTACTS AND LOCATIONS:
Locations (1):
- Médipôle Hôpital Mutualiste, Villeurbanne, France